CLINICAL TRIAL: NCT05959512
Title: A Survey of Smoking Patterns and Influencing Factors Among Hospitalized Patients
Brief Title: Smoking Pattern and Influencing Factors in Hospitalized Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Beijing Normal University (Other)
Responsible Party: Sponsor
Other Study IDs: Smoking pattern in patients
Record Dates: First submitted 2023-07-10; First posted 2023-07-25 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Smoking Behaviors
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study examines the smoking patterns and determinants of inpatients who smoke, develops tailored smoking cessation interventions based on their individual needs, and aims to enhance the effectiveness of quitting and lower the likelihood of relapse.

DETAILED DESCRIPTION:
Smoking is a major risk factor for many chronic and acute diseases, and quitting smoking can bring significant health benefits. However, many smokers find it hard to quit or relapse after quitting. This study aims to explore the smoking behavior and influencing factors of inpatients who smoke. The survey will collect data on the demographic, clinical, psychological, and behavioral aspects of the participants, as well as their smoking history, nicotine dependence, withdrawal symptoms, confidence and motivation to quit, and perceived barriers and facilitators to quitting.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 and above;
2. smoke at least 1 cigarette daily;
3. willing to participate in this study

Exclusion Criteria:

1. Smokers who have mental illness or cognitive impairment;
2. Unable to complete the questionnaire survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of hospitalized patients who smoke and meet the following inclusion and exclusion criteria. Inclusion criteria: (1) Aged 18 years or above; (2) Have a history of smoking, smoking ≥1 cigarette per day (3) Willing to participate in this study and sign an informed consent form. Exclusion criteria: (1) Have mental illness or cognitive impairment; (2) Unable to complete the questionnaire survey.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-07-19 (Actual); Primary Completion 2024-07-14 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Smoking cessation rate at 6 months after discharge | 6 months after discharge
  The number of participants who quit smoking at 6 months after discharge, verified by carbon monoxide (CO) test

SECONDARY OUTCOMES:
Smoking reduction rate at 6 months after discharge | 6 months after discharge
  The number of participants who reduce their daily cigarette consumption by at least 50% at 6 months after discharge
Quit attempt rate during the 6-month follow-up period | 6 months after discharge
  The number of participants who make at least one quit attempt during the 6-month follow-up period, verified by self-report

CONTACTS AND LOCATIONS:
Overall Officials: Xue Weng, Principal Investigator — Beijing Normal University
Locations (1):
- Xue Weng, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: No